CLINICAL TRIAL: NCT01675726
Title: QUALITY OF LIFE OF CHILDREN BORN VERY PRETERM AT SCHOOL-AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A00193-40; 2012-02 (Other: AP HM)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: CHILDREN BORN VERY PRETERM AT SCHOOL-AGE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- quality of life (Other)
  Interventions: Other: questionary on quality of life

INTERVENTIONS:
Other: questionary on quality of life

SUMMARY:
AIMS The aims were 1) to describe the quality of life (QoL) of a cohort of children born very preterm (<28 weeks of gestation) aged 7 to 9 years; 2) to compare children's QoL to the QoL reported by a French general population of reference. 3) to determine whether socio-demographic factors, neonatal features and neurocognitive status were impacting their QoL.

METHODS:

* Multi-centre study: 6 French level three perinatal care units (Marseille, Montpellier, Nantes, Nîmes, Nice and Rouen).
* Inclusion criteria: all infants born before 28 weeks of gestation between January 2005 and December 2007, from 7 to 9 years old of age at the time of evaluation.
* Written agreement to participate: collected from parents.
* Data collection: reports of children's QoL by children and their parents (using standardized validated questionnaires); clinical information about the children, obtained through a medical examination; children neurocognitive profile.
* Duration of inclusion: over 24 months.
* Population: of the six structures, approximately 300 children will be evaluated consistent with the active files of the participating centres and an attrition rate of 30%.

PERSPECTIVES This is one of the first studies to collect self-reported data on quality of life of school-age children (7-9 years) born before 28 weeks of gestation. A better understanding of demographic and clinical determinants of QOL of school-age very preterm children may help clinicians involved in the care of these children in their ethical and medical considerations.

ELIGIBILITY:
Inclusion Criteria:

* Child been born between 01/01/2005 and the inclusive 31/12/2007,
* Extreme premature born Child before 28 weeks of amenorrhea,
* Child hospitalized after the birth in a level maternity 3 (been born " inborn " or " outborn ")
* Not dead Child,
* Child not presenting a cerebral palsy,
* Child capable of answering a questionnaire in French language,
* Child among whom the parents(relatives) or the legal representatives accepted the principle of the participation in this study, and having signed a consent,
* Child granting to participate in the study.

Exclusion Criteria:

* Child died between the birth and dates her(it) evaluation,
* Child presenting a cerebral palsy
* Child among whom the parents(relatives) or the legal representatives refused that their child participates in this study

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
data on quality of life of school-age children born prematurely | 3 years

SECONDARY OUTCOMES:
better understanding of demographic and clinical determinants of QOL of school-age | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Gire C, Resseguier N, Brevaut-Malaty V, Marret S, Cambonie G, Souksi-Medioni I, Muller JB, Garcia P, Berbis J, Tosello B, Auquier P; GPQoL study Group. Quality of life of extremely preterm school-age children without major handicap: a cross-sectional observational study. Arch Dis Child. 2019 Apr;104(4):333-339. doi: 10.1136/archdischild-2018-315046. Epub 2018 Jun 30. PMID 29960997